CLINICAL TRIAL: NCT03082274
Title: Prospective Validation of Prostate Biomarkers for Repeat Biopsy: The PRIORITY Study
Brief Title: Prospective Validation of Prostate Biomarkers for Repeat Biopsy
Acronym: PRIORITY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: MDx Health (Industry)
Responsible Party: Sponsor
Other Study IDs: PRIORITY
Record Dates: First submitted 2017-02-28; First posted 2017-03-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma from each subject will be collected and stored for up to 10 years for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men age 40-85 years with an initial negative prostate biopsy: Men age 40 - 85 years of age Previous negative prostate biopsy within 30 months.
  Interventions: Diagnostic Test: ConfirmMDx; Diagnostic Test: SelectMDx

INTERVENTIONS:
Diagnostic Test: ConfirmMDx — ConfirmMDx is a molecular diagnostic assay which utilizes DNA isolated from biopsy tissues to determine if aberrant DNA methylation is occurring in three genes: GSTP1, RASSF1 and APC. ConfirmMDx is currently available to clinicians for use in cancer-negative extended-core biopsies to determine if occult cancer is present in the prostate.
Diagnostic Test: SelectMDx — SelectMDx for Prostate Cancer is a reverse-transcription PCR (RT-PCR) assay performed on post-DRE, first-void urine specimens from patients with clinical risk factors for prostate cancer, who are being considered for biopsy. The test measures the mRNA levels of the DLX1 and HOXC6 biomarkers, using KLK3 as internal reference gene, to aid in patient selection for prostate biopsy.

SUMMARY:
Target enrollment is 1000 prospectively enrolled subjects with an initial negative biopsy scheduled for repeat biopsy.

Subjects must have had their negative index prostate biopsy procedure within 30 months of being scheduled for their repeat biopsy.

All enrolled subjects will have all core tissues from the initial negative biopsy blinded and tested with the assay.

All subjects will have serum and plasma samples obtained prior to DRE, and a urine sample collected immediately following DRE but in advance of the repeat biopsy; samples will be blinded and sent to MDxHealth for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged 40 years to 85, who underwent a previous cancer-negative prostate biopsy within 30 months of being scheduled for a repeat biopsy.
* The initial TRUS guided negative prostate biopsy must have collected a minimum of 10 tissue cores and sections from all prostate biopsy cores collected by the physician must be submitted to MDxHealth in order to allow for full comprehensive testing/evaluation of all the sections of the patient's prostate prior to the scheduled repeat biopsy.
* Minimum tissue volume criteria of 20 microns of prostate biopsy core tissue is available (40 microns preferable).
* Previous biopsy histology may include the presence of high-grade prostatic intraepithelial neoplasia (HGPIN), proliferative inflammatory atrophy (PIA), glandular inflammation, atypical small acinar proliferation (ASAP) or atypical cells.
* Tissue was extracted using standard TRUS guided biopsy core extraction (and not transurethral resection of the prostate (TURP).
* Pre-DRE serum sample, pre-DRE plasma sample, and Post-DRE urine sample to be collected in advance of the repeat biopsy. Samples can be collected within three months of the scheduled repeat biopsy, up until the day of, but prior to, the procedure.

Exclusion Criteria:

* Patient who has undergone previously testing by ConfirmMDx from the same biopsy
* Patients with prior diagnosis of prostate cancer in any previous biopsy.
* Patients with a limited life expectancy and generally not considered for a repeat Tissue extracted using transurethral resection of the prostate (TURP) procedures
* Patients with a history of cancer (except basal cell carcinoma)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ConfirmMDx assay will be utilized to blindly test the needle biopsy cores of the index negative prostate biopsy (all cores) of men about to undergo repeat prostate biopsy. It is postulated that the test may aid in improved patient risk stratification for repeat biopsy, discriminating patients with no cancer/low grade prostate cancer (GS6) who are at sufficiently low risk to avoid repeat biopsy, while also identifying patients at increased risk for clinical significant disease (≥ GS7) who may benefit from early intervention.
  In this current study, SelectMDx will be used to blindly test urine samples obtained preceding a repeat prostate biopsy to validate the test's ability to predict risk for high-grade disease. The intent is to demonstrate the test's ability to non-invasively stratify those patients at risk for aggressive disease, who require a repeat prostate biopsy, versus those at sufficiently low risk who may avoid unnecessary repeat biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Validate ConfirmMDx for Prostate Cancer to predict the outcome of repeat biopsy | 1 year
  The primary objectives of this prospective, multi-center study are twofold:
  * Validate use of the ConfirmMDx for Prostate Cancer to predict the outcome of a repeat biopsy in men with a previous negative prostate biopsy using tissue.
  * Validate use of the SelectMDx for Prostate Cancer to predict the outcome of a repeat biopsy in men with a previous negative prostate biopsy using urine.

SECONDARY OUTCOMES:
Comparison between clinical and pathological outcomes | 1 year
  Subset analyses conducted in appropriate groups, such as patients with available data from radical prostatectomy, and correlate this data with the ConfirmMDx and SelectMDx results.
  * Evaluate rate of cancer detection on repeat biopsy and associated complications.
  * Evaluate the findings of MRI fusion biopsy with standard 12 core TRUS guided biopsy (if available).

CONTACTS AND LOCATIONS:
Locations (1):
- MDxHealth, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No